CLINICAL TRIAL: NCT03527121
Title: Management of Acute Lateral Ankle Sprains: A Randomized Controlled Trial
Brief Title: Management of Acute Lateral Ankle Sprains
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Christian Olsen (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other); Regionshospitalet Horsens (Other); University of Copenhagen (Other); Slagelse Hospital (Other)
Responsible Party: Sponsor-Investigator, Christian Olsen, Principal Investigator, Slagelse Hospital
Organization: Slagelse Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SJ-628
Record Dates: First submitted 2018-04-24; First posted 2018-05-17 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Ankle Sprains
Keywords: Ankle; Exercise; Activities of daily living; Treatment outcome
MeSH Terms: conditions — Ankle Injuries; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R.I.C.E.+ (ESP physiotherapy) (Experimental): Participants will receive a single session with advice and instructions from an ESP physiotherapist in rest, ice, compression and elevation AND pain guided early weight bearing plus a written home-based exercise program.
  Interventions: Other: ESP physiotherapy
- R.I.C.E.(Usual care) (Active Comparator): A single session with advice and instructions from a physician in rest, ice, compression and elevation.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: ESP physiotherapy — A single session with advice and instructions from an ESP physiotherapist in rest, ice, compression and elevation AND pain guided early weight bearing plus a written home-based exercise program.
  Arms: R.I.C.E.+ (ESP physiotherapy)
Other: Usual care — A single session with advice and instructions from a physician in rest, ice, compression and elevation (usual care group).
  Arms: R.I.C.E.(Usual care)

SUMMARY:
This study evaluates the effectiveness of pain guided early weight bearing as a means to enhance the outcome of acute lateral ankle sprain. Half of the participants will receive advice and instructions in pain guided early weight bearing plus a written home-based exercise program, while the other half will receive advice and instructions following standard operating procedures at site.

DETAILED DESCRIPTION:
Lateral ankle sprains (LAS) is the most common injury in the active population. Not only is the injury prevalent within organized sports, but also display high prevalence in the general population presenting at the emergency departments (ED). LAS accounts for about 3-5% of all visits to the ED, but total LAS incidence rates are increasing in the general population.

Acute LAS is defined by Delahunt et al. and endorsed by the International ankle consortium as: "An acute traumatic injury to the lateral ligament complex of the ankle joint as a result of excessive inversion of the rear foot or a combined plantar flexion and adduction of the foot." The treatment of LAS in the emergency department consists of initial assessment and acute management of the injured foot, traditionally done by a physician. The typical assessment consists of ruling out severe injury, i.e. fracture, using the Ottawa ankle foot rules. The acute management of the injured ankle is typically composed of a treatment approach consisting of Rest, Ice, Compression and Elevation (RICE).

Extended Scope of Practice (ESP) physiotherapists in EDs have shown to generate high levels of patient satisfaction, reduce patient waiting times and have high clinical effectiveness, yet high quality randomized trials investigating the clinically effectiveness of ESP physiotherapy are lacking. Acute LAS is one of the most common injuries managed in EDs and poor functional status within the initial 2 weeks after injury is predictive of development of chronic ankle instability (CAI), which can be a serious barrier for future physical activity and occupational performance. Early and targeted interventions provided in the emergency department by ESP physiotherapists may therefore prove to be beneficial for the patients and the society.

The aim of this RCT is to investigate if pain guided early weight bearing provided by ESP physiotherapists is superior to advice and instructions following standard operating procedures provided by a physician in improving the selfreported functional outcome in patients with LAS.

The study hypothesis is that patients randomized to pain guided early weight bearing will improve significantly more in the lower extremity functional scale after 4 weeks than those randomized to standard care.

ELIGIBILITY:
Inclusion Criteria:

1. A grade 1 or 2 LAS sustained within 24 hours of randomization
2. To be a minimum age of 18
3. Signed informed consent

Exclusion Criteria:

1. A grade 3 LAS injury sustained
2. Diagnosed with chronic ankle instability (CAI) on the affected limb
3. Fracture diagnosed by X-ray
4. Previous enrollment in the same study
5. Major lower limb surgery or other severe lower extremity injury in the past 3 months on the affected limb
6. Under the influence of drugs or alcohol
7. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., not having access to the internet, immobilization etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Lower extremity functional scale | Primary endpoint: The change from baseline to 4 weeks. Secondary outcomes: The change from baseline to 1, 2 and 3 weeks, and 3, 6 and 12 months.
  The Lower extremity functional scale is a self-completed questionnaire providing a total score based on the patients subjective ankle function. The scale consists of 20 functional leg activities, each scored on a five point scale (0 impossible, 4 no difficulty), giving a minimum score of 0 (worst) to 80 (best). The questionnaire will be translated into Danish using a dual-panel approach before trial start. The LEFS will be scored online by the trial participant. This approach avoids the requirement for follow-up visits in a clinic.

SECONDARY OUTCOMES:
Foot and ankle ability measure (FAAM) | Primary endpoint: The change from 1 to 4 weeks. Secondary outcomes: The change from 1. week to 2. and 3. weeks, and 3, 6 and 12 months
  The Foot and ankle Ability Measure is a 29-item region-specific outcome instrument. The FAAM ADL subscale consist of 21-items and the FAAM sports consist of 8-items. Each item is scored on a 5-point Likert scale (4 to 0) from 'no difficulty at all' to 'unable to do'. N/A responses are not counted. Item total scores range from 0 to 84 for the ADL subscale and 0 to 32 for the Sports subscale, with higher scores representing better function. For both subscales, the score on each item are added together to get the item score total. The number of items with a response is multiplied by 4 to get the highest potential score. The item score total is divided by the highest potential score. This value is multiplied by 100 to get a final percentage score. Evidence of validity to support the use of the FAAMadl and FAAMsport is available in individuals with a wide array of ankle and foot disorders. The questionnaire will be translated into Danish using a dual-panel approach before trial start.
Reinjury rates | Primary endpoint: The difference in reinjury from baseline to 4 weeks. Secondary outcomes: 2 and 3 weeks, and 3, 6 and 12 months
  The investigators endorse the definition of an ankle sprain as: "An acute traumatic injury to the lateral ligament complex of the ankle joint as a result of excessive inversion of the rear foot or a combined plantar flexion and adduction of the foot. This usually results in some initial deficits of function and disability". Reinjury will not be considered as a stopping rule for further participation in this study.
Global perceived effect (GPE) | Primary endpoint: After 4 weeks. Secondary outcomes: 1, 2 and 3 weeks, and 3, 6 and 12 months.
  Perceived effect of treatment will be measured using a transition questionnaire (TRANS-Q) on which the participants will answer if their current LAS-related health status is "unchanged", "worse" or "better" compared to their pre-LAS status. An "unchanged" equals a transition score of 0. If the participant answers "worse", he/she is asked to rate the degree of worsening on a 7 point Likert scale, and the corresponding scores range from -1 to -7. If a participant answers "better", he/she is asked to rate the degree of improvement on a 7 point Likert scale, and the corresponding scores range from 1 to 7.
Adverse events (AE) and serious adverse events (SAE) | Recorded at all follow-ups: 1, 2, 3 and 4 weeks and 3, 6 and 12 months
  Adverse events (AE) and serious adverse events (SAE) will be recorded at all follow-ups by asking the participants about potential AEs using open-probe questioning to ensure that all AEs are recorded. AEs will be categorized into index foot or other sites and will be recorded and assessed for severity independent of whether or not there is a causal relationship with study treatments.

OTHER OUTCOMES:
Pain at rest and with activity, assessed using a visual analogue scale (VAS) | Primary endpoint: The change from baseline to 4 weeks. Secondary outcomes: 1, 2 and 3 weeks, and 3, 6 and 12 months.
  The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations. The scale is a continuous scale comprised of a horizontal line, anchored by 2 verbal descriptors, one for each symptom extreme (0 no pain, 10 the worst imaginable pain). We will measure pain VAS at rest and pain VAS with activity.
The Cumberland ankle instability tool (CAIT) | Primary endpoint: The change from baseline to 4 weeks. Secondary outcomes: 1, 2 and 3 weeks, and 3, 6 and 12 months.
  The CAIT is a simple, validated, and reliable tool to measure severity of functional ankle instability. The CAIT consists of 9 questions that are answered separately for the right and left ankle. It is scored on a 30-point scale, with lower scores indicating decreased stability. The minimal clinically important difference (MCID) for patients with chronic ankle instability is ≥3 points.
Quality of life (EQ-5D-3L) | Primary endpoint: The change from baseline to 4 weeks. Secondary outcomes: 1, 2 and 3 weeks, and 3, 6 and 12 months.
  The EQ-5D-3L is a measure of current health status developed by the EuroQol Group for clinical and economic appraisals. The questionnaire consists of five questions assessing five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension is rated on three levels: no problems, some problems and extreme problems.
Patient acceptable symptom state (PASS) | Primary endpoint: The change from baseline to 4 weeks. Secondary outcomes: 1, 2 and 3 weeks, and 3, 6 and 12 months.
  The PASS is the value beyond which patients consider themselves well. Patients' opinions of their state will be recorded by answering ''Yes'' or ''No'' to the question: ''Taking into account all the activities you have during your daily life, your level of pain, and also your functional impairment, do you consider your current state is satisfactory?''.
Patient-reported treatment failure | Primary endpoint: The change from baseline to 4 weeks. Secondary outcomes: 1, 2 and 3 weeks, and 3, 6 and 12 months.
  Only answered by patients answering "no" to PASS. "Would you consider your current state as being so unsatisfactory that you consider the treatment to have failed?". Answered by "yes" or "no".
Analgesic use | Primary endpoint: The change from 1. to 4. week. Secondary outcomes: The change from week 1. to 2. and 3. weeks.
  The participants self-reported use of analgesics will be collected at baseline and at follow-up week 1, 2, 3 and 4. Participants will be asked to note their use of analgesic drugs within the week before baseline and the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Christian P Olsen, PT, Msc, Principal Investigator — Department of Physiotherapy and Occupational Therapy, Slagelse Hospitals.; Marius Henriksen, PT, Prof., Study Chair — University of Copenhagen and Bispebjerg-Frederiksberg Hospital; Søren T Skou, PT, PhD, Study Chair — University of Southern Denmark and Naestved-Slagelse-Ringsted Hospitals.; Mikael Elsborg, PT, Study Chair — The Regional Hospital in Horsens
Locations (2):
- Denmark (2):
  - The Emergency Department, Slagelse Hospital, Slagelse, Region Sjælland
  - The Emergency Department, The Regional Hospital in Horsens, Horsens, The Central Region of Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT03527121/Prot_SAP_ICF_000.pdf